CLINICAL TRIAL: NCT04910425
Title: Phase II Study to Evaluate the Performance of PSMA-Targeted 18F-DCFPyL PET/MRI for the Detection of Clinically Significant Prostate Cancer in Men Presenting Following a Positive Screen for Prostate Cancer
Brief Title: PSMA-Targeted 18F-DCFPyL PET/MRI for the Detection of Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study aborted
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NU 19U05; NCI-2021-05593 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00212326; NU 19U05 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid; gadobenic acid; gadobutrol; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (18F-DCFPyL PET/MRI, mpMRI) (Experimental): Patients receive fluorine F 18 DCFPyL IV and undergo PET/MRI. Patients also receive either gadobutrol IV or gadobenate dimeglumine IV (per radiologist preference), and undergo mpMRI. Within approximately 60 days after PET/MRI and mpMRI, patients undergo TRUS guided prostate biopsy per standard of care.
  Interventions: Drug: Fluorine F 18 DCFPyL; Drug: Gadobenate Dimeglumine; Drug: Gadobutrol; Procedure: Magnetic Resonance Imaging; Procedure: Multiparametric Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Transrectal Ultrasonography Guided Biopsy

INTERVENTIONS:
Drug: Fluorine F 18 DCFPyL — Given IV
  Other Names: 18F-DCFPyL
Drug: Gadobenate Dimeglumine — Given IV
  Other Names: Gd-BOPTA; MultiHance
Drug: Gadobutrol — Given IV
  Other Names: BAY86-4875; Gadavist; Gadograf; Gadovist; Protovis; ZK 135079
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Multiparametric Magnetic Resonance Imaging — Undergo mpMRI
  Other Names: MP-MRI; mpMRI; Multi-parametric MRI; Multiparametric MRI
Procedure: Positron Emission Tomography — Undergo PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Procedure: Transrectal Ultrasonography Guided Biopsy — Undergo TRUS-guided biopsy
  Other Names: TRUS Biopsy; TRUS-Guided Biopsy

SUMMARY:
This phase II trial studies how well 18F-DCFPyL positron emission tomography (PET)/magnetic resonance imaging (MRI) works for the diagnosis of prostate cancer in men with a PSA greater than or equal to 2 ng/mL. 18F-DCFPyl is a radioactive injectable imaging agent made of a prostate specific membrane antigen (PSMA) that attaches to tumor cells, which makes it useful for the diagnosis of prostate cancer. A PET scan is an imaging tool that may help find the location of cancer, by using a radioactive drug and a computer to create images of how organs and tissues in the body are functioning. A mp-MRI is used to help determine the extent of a patient's cancer. A MRI scan uses strong magnets and computers to create detailed images of the soft tissue in the body. This trial aims to compare PET scans to prostate specific mp-MRI to evaluate prostate cancer severity in men with a positive screen for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare the fluorine F 18 DCFPyL (18-F-DCFPyL) PET to multiparametric magnetic resonance imaging (mpMRI) for the diagnosis of clinically significant prostate cancer in biopsy naive men as defined by Gleason score >= 3+4 (International Society of Urological Pathology [ISUP] group >= 2).

SECONDARY OBJECTIVES:

I. Compare the combined 18-F-DCFPyL PET and mpMRI to mpMRI alone for the diagnosis of clinically significant prostate cancer in biopsy naive men as defined by Gleason score >= 3+4 (ISUP group >= 2).

II. Estimate the sensitivities and specificities of combined 18-F-DCFPyL PET/mpMRI, mpMRI alone, 18-F-DCFPyL PET alone, and prostate health index (PHI) alone for the diagnosis of clinically significant prostate cancer.

III. Estimate the accuracy of PET alone for the diagnosis of clinically significant prostate cancer in biopsy naïve men as defined by Gleason score >= 3+4 (ISUP group >=2).

IV. Compare the accuracy of PET to prostate health index (PHI) for the diagnosis of clinically significant prostate cancer in biopsy naive men as defined by Gleason score >= 3+4 (ISUP group >= 2).

OUTLINE:

Patients receive fluorine F 18 DCFPyL intravenously (IV) and undergo PET/MRI. Patients also receive either gadobutrol IV or gadobenate dimeglumine IV (per radiologist preference), and undergo mpMRI. Within approximately 60 days after PET/MRI and mpMRI, patients undergo transrectal ultrasound (TRUS) guided prostate biopsy per standard of care.

After completion of study intervention, patients are followed up within 24 hours, and then at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a positive screen for prostate cancer as confirmed by a prostate specific antigen (PSA) >= 2 ng/ml
* Patients must elect to elect to undergo PHI blood test and TRUS-guided elect to undergo PHI blood test and TRUS-guided biopsy as part of routine clinical care
* Patients must be age >= 18 years
* Patients must agree to use adequate contraception (e.g. Barrier method of birth control; abstinence) for 24 hours following completion of imaging
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Patients who have had a prior biopsy for prostate cancer
* Patients who have contraindications to MRI (i.e. pacemakers, aneurysm clips or shaped fragments) are not eligible
* Patients receiving any other treatments or investigational agents are not eligible
* Patients with a glomerular filtration rate (GFR) < 30mL/min are ineligible to receive intravenous contrast per standard magnetic resonance (MR) exclusion criteria
* Patients administered a radioisotope < 5 physical half-lives prior to the date of study PET/MRI
* Patients administered IV X-ray contrast medium < 120 hours prior to the date of study PET/MRI
* Patients who report taking multivitamins on the day of study PET/MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-17 (Estimated); Primary Completion 2026-06-17 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
18-F-DCFPyL positron emission tomography (PET) vs multiparametric magnetic resonance imaging (mpMRI) for the diagnosis of clinically significant prostate cancer in biopsy naïve men. | Up to 30 days
  Will be compared to multiparametric magnetic resonance imaging (mpMRI) for the diagnosis of clinically significant prostate cancer in biopsy naive men as defined by Gleason score >= 3+4 (International Society of Urological Pathology [ISUP] group >=2).

SECONDARY OUTCOMES:
Sensitivity of combined PET-mpMRI to mpMRI | Up to 30 days
  Will be estimated and compared to mpMRI alone for the diagnosis of clinically significant prostate cancer in biopsy naive men as defined by Gleason score >= 3+4 (ISUP group >= 2).

CONTACTS AND LOCATIONS:
Overall Officials: Edward M Schaeffer, MD/PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States